CLINICAL TRIAL: NCT00063063
Title: Generic Database: A Survey of Morbidity and Mortality in Very Low Birth Weight Infants
Brief Title: Generic Database of Very Low Birth Weight Infants
Acronym: GDB
Status: Recruiting | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-NRN-0001; U24HD095254 (NIH); UG1HD068263 (NIH); UG1HD034216 (NIH); UG1HD021364 (NIH); UG1HD027853 (NIH); UG1HD027851 (NIH); UG1HD053109 (NIH); UG1HD112079 (NIH); UG1HD112093 (NIH); UG1HD027904 (NIH); UG1HD053089 (NIH); UG1HD068244 (NIH); UG1HD027880 (NIH); UG1HD087226 (NIH); UG1HD040689 (NIH); UG1HD040492 (NIH); UG1HD112097 (NIH); UG1HD112100 (NIH); UG1HD068278 (NIH)
Record Dates: First submitted 2003-06-19; First posted 2003-06-20 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Registry Cohort: Registry Cohort
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
The Generic Database (GDB) is a registry of very low birth weight infants born alive in NICHD Neonatal Research Network (NRN) centers. The GDB collects observational baseline data on both mothers and infants, and the therapies used and outcomes of the infants. The information collected is not specific to a disease or treatment (i.e., it is "generic"). Data are analyzed to find associations and trends between baseline information, treatments, and infant outcome, and to develop future NRN trials.

DETAILED DESCRIPTION:
The Generic Database (GDB) is a registry of very low birth weight infants born alive in NICHD Neonatal Research Network (NRN) centers. The purpose is to collect baseline and outcome data in a uniform manner on a large cohort of VLBW and other sick infants admitted to neonatal intensive care units.

The GDB collects observational baseline data on both mothers and infants, and the therapies used and outcomes of the infants. The information collected is not specific to a disease or treatment (i.e., it is "generic"). Baseline data is collected soon after admission to the NICU; outcome data is collected at the time of death or discharge from the hospital. The data collected includes information on:

* Demographics of mother and infant
* Mother's health (e.g., pregnancy history and complications)
* Labor and deliver (e.g., rupture of the membranes, steroids and antibiotics given, mode of delivery)
* Infant's health (gestational age, Apgar scores, weight, length, delivery room resuscitation, respiratory support, etc.)
* Infant's medical outcome (heart, lung, nervous system, gastrointestinal system, hearing, and vision, known infections, and major malformations/syndromes, and mortality or number of days hospitalized).

These data are used: to examine associations between baseline characteristics, treatments, and outcomes; to track trends in incidences of disease and effectiveness of therapies; and to identify questions requiring additional in-depth research.

Informed Consent: As required by local IRBs.

Secondary Studies include:

A. The All Birth Cohort (ABC) Study. A time-limited observational registry to determine the incidence of intrapartum stillbirth at 20 0/7 - 28 6/7 weeks' gestation and its associated factors at Network sites.

ELIGIBILITY:
Inclusion Criteria:

* Infants inborn at NICHD NRN centers that are:
* 401-1000 grams birth weight, and/or
* 20 0/7 to 28 6/7 weeks (<29 weeks) gestational age
* Infants enrolled in one or more additional NICHD NRN interventional trials or time-limited observational studies. For infants that do not meet the inclusion criteria above, inclusion and exclusion criteria for the Generic Database are determined by the criteria for the additional trial(s). In these cases, infants that are larger than 1,000 grams and/or older than 29 weeks may be included in the GDB.

Exclusion Criteria:

* Infants >1,000 grams birth weight and/or >29 weeks gestational age

Note: These inclusion criteria were changed as of 1/1/2008. Prior to this date, all infants with birth weights between 401 and 1500 grams who are admitted to NRN NICUs within 14 days of birth were included in the database.

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants inborn at NICHD NRN centers that are 401-1000 grams birth weight, and/or <29 weeks gestational age, OR infants enrolled in one or more additional NICHD NRN studies.
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 1987-04-01 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
To maintain a registry of baseline and outcome data for VLBW infants with data collected in a uniform manner | Longitudinal database currently funded through 3/31/2030
  To maintain a registry of baseline and outcome data for VLBW infants with data collected

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Anna Maria Hibbs, MD, MSCE, FAAP, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; C. Michael Cotten, MD, Principal Investigator — Duke University; Ravi M Patel, MD, MSc, Study Chair — Emory University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P Van Meurs, MD, Principal Investigator — Stanford University; Stephanie Merhar, MD MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Tarah Colaizy, MD, MPH, Principal Investigator — University of Iowa; Kristi L Watterberg, MD, Principal Investigator — University of New Mexico; Myra Wyckoff, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Jon E Tyson, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Sara DeMauro, MD, MSCE, Principal Investigator — University of Pennsylvania; Carl D'Angio, MD, Principal Investigator — University of Rochester; Pablo Sanchez, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital; Robin Ohls, MD, Principal Investigator — University of Utah
Locations (31):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California at San Diego, San Diego, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Harvard University, Cambridge, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of Mississippi Medical Center - Children's of Mississippi, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Background] Strand M, Jobe AH. The multiple negative randomized controlled trials in perinatology--why? Semin Perinatol. 2003 Aug;27(4):343-50. doi: 10.1016/s0146-0005(03)00042-9. PMID 14510325
- [Background] Tyson JE, Stoll BJ. Evidence-based ethics and the care and outcome of extremely premature infants. Clin Perinatol. 2003 Jun;30(2):363-87. doi: 10.1016/s0095-5108(03)00028-9. PMID 12875360
- [Background] Wright LL. How to develop and manage a successful research network. Semin Pediatr Surg. 2002 Aug;11(3):175-80; discussion 180. doi: 10.1053/spsu.2002.33740. No abstract available. PMID 12145760
- [Background] Wright LL, McNellis D. National Institute of Child Health and Human Development (NICHD)-sponsored Perinatal Research Networks. Semin Perinatol. 1995 Apr;19(2):112-23. doi: 10.1016/s0146-0005(05)80031-x. No abstract available. PMID 7604302
- [Result] Adams-Chapman I, Hansen NI, Stoll BJ, Higgins R; NICHD Research Network. Neurodevelopmental outcome of extremely low birth weight infants with posthemorrhagic hydrocephalus requiring shunt insertion. Pediatrics. 2008 May;121(5):e1167-77. doi: 10.1542/peds.2007-0423. Epub 2008 Apr 7. PMID 18390958
- [Result] Ambalavanan N, Carlo WA, Bobashev G, Mathias E, Liu B, Poole K, Fanaroff AA, Stoll BJ, Ehrenkranz R, Wright LL; National Institute of Child Health and Human Development Neonatal Research Network. Prediction of death for extremely low birth weight neonates. Pediatrics. 2005 Dec;116(6):1367-73. doi: 10.1542/peds.2004-2099. PMID 16322160
- [Result] Benjamin DK Jr, Stoll BJ, Fanaroff AA, McDonald SA, Oh W, Higgins RD, Duara S, Poole K, Laptook A, Goldberg R; National Institute of Child Health and Human Development Neonatal Research Network. Neonatal candidiasis among extremely low birth weight infants: risk factors, mortality rates, and neurodevelopmental outcomes at 18 to 22 months. Pediatrics. 2006 Jan;117(1):84-92. doi: 10.1542/peds.2004-2292. PMID 16396864
- [Result] Broitman E, Ambalavanan N, Higgins RD, Vohr BR, Das A, Bhaskar B, Murray K, Hintz SR, Carlo WA; National Institute of Child Health and Human Development Neonatal Research Network. Clinical data predict neurodevelopmental outcome better than head ultrasound in extremely low birth weight infants. J Pediatr. 2007 Nov;151(5):500-5, 505.e1-2. doi: 10.1016/j.jpeds.2007.04.013. Epub 2007 Jul 12. PMID 17961693
- [Result] Castro L, Yolton K, Haberman B, Roberto N, Hansen NI, Ambalavanan N, Vohr BR, Donovan EF. Bias in reported neurodevelopmental outcomes among extremely low birth weight survivors. Pediatrics. 2004 Aug;114(2):404-10. doi: 10.1542/peds.114.2.404. PMID 15286223
- [Result] Cole CR, Hansen NI, Higgins RD, Ziegler TR, Stoll BJ; Eunice Kennedy Shriver NICHD Neonatal Research Network. Very low birth weight preterm infants with surgical short bowel syndrome: incidence, morbidity and mortality, and growth outcomes at 18 to 22 months. Pediatrics. 2008 Sep;122(3):e573-82. doi: 10.1542/peds.2007-3449. PMID 18762491
- [Result] Cotten CM, Oh W, McDonald S, Carlo W, Fanaroff AA, Duara S, Stoll B, Laptook A, Poole K, Wright LL, Goldberg RN; NICHD Neonatal Research Network. Prolonged hospital stay for extremely premature infants: risk factors, center differences, and the impact of mortality on selecting a best-performing center. J Perinatol. 2005 Oct;25(10):650-5. doi: 10.1038/sj.jp.7211369. PMID 16079906
- [Result] Cotten CM, Taylor S, Stoll B, Goldberg RN, Hansen NI, Sanchez PJ, Ambalavanan N, Benjamin DK Jr; NICHD Neonatal Research Network. Prolonged duration of initial empirical antibiotic treatment is associated with increased rates of necrotizing enterocolitis and death for extremely low birth weight infants. Pediatrics. 2009 Jan;123(1):58-66. doi: 10.1542/peds.2007-3423. PMID 19117861
- [Result] Da Costa D, Bann CM, Hansen NI, Shankaran S, Delaney-Black V; National Institute of Child Health and Human Development Neonatal Research Network. Validation of the Functional Status II questionnaire in the assessment of extremely-low-birthweight infants. Dev Med Child Neurol. 2009 Jul;51(7):536-44. doi: 10.1111/j.1469-8749.2009.03318.x. PMID 19459909
- [Result] Demarini S, Dollberg S, Hoath SB, Ho M, Donovan EF. Effects of antenatal corticosteroids on blood pressure in very low birth weight infants during the first 24 hours of life. J Perinatol. 1999 Sep;19(6 Pt 1):419-25. doi: 10.1038/sj.jp.7200245. PMID 10685271
- [Result] Dollberg S, Demarini S, Donovan EF, Hoath SB. Maturation of thermal capabilities in preterm infants. Am J Perinatol. 2000;17(1):47-51. doi: 10.1055/s-2000-7293. PMID 10928604
- [Result] Donovan EF, Ehrenkranz RA, Shankaran S, Stevenson DK, Wright LL, Younes N, Fanaroff AA, Korones SB, Stoll BJ, Tyson JE, Bauer CR, Lemons JA, Oh W, Papile LA. Outcomes of very low birth weight twins cared for in the National Institute of Child Health and Human Development Neonatal Research Network's intensive care units. Am J Obstet Gynecol. 1998 Sep;179(3 Pt 1):742-9. doi: 10.1016/s0002-9378(98)70075-4. PMID 9757982
- [Result] Doyle NM, Gardner MO, Wells L, Qualls C, Papile LA. Outcome of very low birth weight infants exposed to antenatal indomethacin for tocolysis. J Perinatol. 2005 May;25(5):336-40. doi: 10.1038/sj.jp.7211256. PMID 15861198
- [Result] Ehrenkranz RA, Walsh MC, Vohr BR, Jobe AH, Wright LL, Fanaroff AA, Wrage LA, Poole K; National Institutes of Child Health and Human Development Neonatal Research Network. Validation of the National Institutes of Health consensus definition of bronchopulmonary dysplasia. Pediatrics. 2005 Dec;116(6):1353-60. doi: 10.1542/peds.2005-0249. PMID 16322158
- [Result] Ehrenkranz RA, Wright LL. NICHD neonatal research network: contributions and future challenges. Semin Perinatol. 2003 Aug;27(4):264-80. doi: 10.1016/s0146-0005(03)00041-7. PMID 14510317
- [Result] Fanaroff AA, Hack M, Walsh MC. The NICHD neonatal research network: changes in practice and outcomes during the first 15 years. Semin Perinatol. 2003 Aug;27(4):281-7. doi: 10.1016/s0146-0005(03)00055-7. PMID 14510318
- [Result] Fanaroff AA, Stoll BJ, Wright LL, Carlo WA, Ehrenkranz RA, Stark AR, Bauer CR, Donovan EF, Korones SB, Laptook AR, Lemons JA, Oh W, Papile LA, Shankaran S, Stevenson DK, Tyson JE, Poole WK; NICHD Neonatal Research Network. Trends in neonatal morbidity and mortality for very low birthweight infants. Am J Obstet Gynecol. 2007 Feb;196(2):147.e1-8. doi: 10.1016/j.ajog.2006.09.014. PMID 17306659
- [Result] Fanaroff AA, Wright LL, Stevenson DK, Shankaran S, Donovan EF, Ehrenkranz RA, Younes N, Korones SB, Stoll BJ, Tyson JE, et al. Very-low-birth-weight outcomes of the National Institute of Child Health and Human Development Neonatal Research Network, May 1991 through December 1992. Am J Obstet Gynecol. 1995 Nov;173(5):1423-31. doi: 10.1016/0002-9378(95)90628-2. PMID 7503180
- [Result] Gardner MO, Papile LA, Wright LL. Antenatal corticosteroids in pregnancies complicated by preterm premature rupture of membranes. Obstet Gynecol. 1997 Nov;90(5):851-3. doi: 10.1016/S0029-7844(97)00404-3. PMID 9351778
- [Result] Gargus RA, Vohr BR, Tyson JE, High P, Higgins RD, Wrage LA, Poole K. Unimpaired outcomes for extremely low birth weight infants at 18 to 22 months. Pediatrics. 2009 Jul;124(1):112-21. doi: 10.1542/peds.2008-2742. PMID 19564290
- [Result] Guillet R, Stoll BJ, Cotten CM, Gantz M, McDonald S, Poole WK, Phelps DL; National Institute of Child Health and Human Development Neonatal Research Network. Association of H2-blocker therapy and higher incidence of necrotizing enterocolitis in very low birth weight infants. Pediatrics. 2006 Feb;117(2):e137-42. doi: 10.1542/peds.2005-1543. Epub 2006 Jan 3. PMID 16390920
- [Result] Hack M, Horbar JD, Malloy MH, Tyson JE, Wright E, Wright L. Very low birth weight outcomes of the National Institute of Child Health and Human Development Neonatal Network. Pediatrics. 1991 May;87(5):587-97. PMID 2020502
- [Result] Hack M, Wright LL, Shankaran S, Tyson JE, Horbar JD, Bauer CR, Younes N. Very-low-birth-weight outcomes of the National Institute of Child Health and Human Development Neonatal Network, November 1989 to October 1990. Am J Obstet Gynecol. 1995 Feb;172(2 Pt 1):457-64. doi: 10.1016/0002-9378(95)90557-x. PMID 7856670
- [Result] Heller CD, O'Shea M, Yao Q, Langer J, Ehrenkranz RA, Phelps DL, Poole WK, Stoll B, Duara S, Oh W, Lemons J, Poindexter B; NICHD Neonatal Research Network. Human milk intake and retinopathy of prematurity in extremely low birth weight infants. Pediatrics. 2007 Jul;120(1):1-9. doi: 10.1542/peds.2006-1465. PMID 17606555
- [Result] Hintz SR, Kendrick DE, Vohr BR, Poole WK, Higgins RD; National Institute of Child Health and Human Development (NICHD) Neonatal Research Network. Community supports after surviving extremely low-birth-weight, extremely preterm birth: special outpatient services in early childhood. Arch Pediatr Adolesc Med. 2008 Aug;162(8):748-55. doi: 10.1001/archpedi.162.8.748. PMID 18678807
- [Result] Hintz SR, Bann CM, Ambalavanan N, Cotten CM, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Predicting time to hospital discharge for extremely preterm infants. Pediatrics. 2010 Jan;125(1):e146-54. doi: 10.1542/peds.2009-0810. Epub 2009 Dec 14. PMID 20008430
- [Result] Hintz SR, Kendrick DE, Stoll BJ, Vohr BR, Fanaroff AA, Donovan EF, Poole WK, Blakely ML, Wright L, Higgins R; NICHD Neonatal Research Network. Neurodevelopmental and growth outcomes of extremely low birth weight infants after necrotizing enterocolitis. Pediatrics. 2005 Mar;115(3):696-703. doi: 10.1542/peds.2004-0569. PMID 15741374
- [Result] Hintz SR, Kendrick DE, Vohr BR, Poole WK, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Changes in neurodevelopmental outcomes at 18 to 22 months' corrected age among infants of less than 25 weeks' gestational age born in 1993-1999. Pediatrics. 2005 Jun;115(6):1645-51. doi: 10.1542/peds.2004-2215. PMID 15930228
- [Result] Hintz SR, Kendrick DE, Vohr BR, Kenneth Poole W, Higgins RD; Nichd Neonatal Research Network. Gender differences in neurodevelopmental outcomes among extremely preterm, extremely-low-birthweight infants. Acta Paediatr. 2006 Oct;95(10):1239-48. doi: 10.1080/08035250600599727. PMID 16982497
- [Result] Hintz SR, Poole WK, Wright LL, Fanaroff AA, Kendrick DE, Laptook AR, Goldberg R, Duara S, Stoll BJ, Oh W; NICHD Neonatal Research Network. Changes in mortality and morbidities among infants born at less than 25 weeks during the post-surfactant era. Arch Dis Child Fetal Neonatal Ed. 2005 Mar;90(2):F128-33. doi: 10.1136/adc.2003.046268. PMID 15724036
- [Result] Horbar JD, Onstad L, Wright E. Predicting mortality risk for infants weighing 501 to 1500 grams at birth: a National Institutes of Health Neonatal Research Network report. Crit Care Med. 1993 Jan;21(1):12-8. doi: 10.1097/00003246-199301000-00008. PMID 8420718
- [Result] Horbar JD, Wright EC, Onstad L. Decreasing mortality associated with the introduction of surfactant therapy: an observational study of neonates weighing 601 to 1300 grams at birth. The Members of the National Institute of Child Health and Human Development Neonatal Research Network. Pediatrics. 1993 Aug;92(2):191-6. PMID 7710456
- [Result] Lainwala S, Perritt R, Poole K, Vohr B; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental and growth outcomes of extremely low birth weight infants who are transferred from neonatal intensive care units to level I or II nurseries. Pediatrics. 2007 May;119(5):e1079-87. doi: 10.1542/peds.2006-0899. Epub 2007 Apr 2. PMID 17403821
- [Result] Laptook AR, O'Shea TM, Shankaran S, Bhaskar B; NICHD Neonatal Network. Adverse neurodevelopmental outcomes among extremely low birth weight infants with a normal head ultrasound: prevalence and antecedents. Pediatrics. 2005 Mar;115(3):673-80. doi: 10.1542/peds.2004-0667. PMID 15741371
- [Result] Laptook AR, Salhab W, Bhaskar B; Neonatal Research Network. Admission temperature of low birth weight infants: predictors and associated morbidities. Pediatrics. 2007 Mar;119(3):e643-9. doi: 10.1542/peds.2006-0943. Epub 2007 Feb 12. PMID 17296783
- [Result] Lemons JA, Bauer CR, Oh W, Korones SB, Papile LA, Stoll BJ, Verter J, Temprosa M, Wright LL, Ehrenkranz RA, Fanaroff AA, Stark A, Carlo W, Tyson JE, Donovan EF, Shankaran S, Stevenson DK. Very low birth weight outcomes of the National Institute of Child health and human development neonatal research network, January 1995 through December 1996. NICHD Neonatal Research Network. Pediatrics. 2001 Jan;107(1):E1. doi: 10.1542/peds.107.1.e1. PMID 11134465
- [Result] Lowe J, Woodward B, Papile LA. Emotional regulation and its impact on development in extremely low birth weight infants. J Dev Behav Pediatr. 2005 Jun;26(3):209-13. doi: 10.1097/00004703-200506000-00008. PMID 15956871
- [Result] Madan JC, Kendrick D, Hagadorn JI, Frantz ID 3rd; National Institute of Child Health and Human Development Neonatal Research Network. Patent ductus arteriosus therapy: impact on neonatal and 18-month outcome. Pediatrics. 2009 Feb;123(2):674-81. doi: 10.1542/peds.2007-2781. PMID 19171637
- [Result] Malcolm WF, Gantz M, Martin RJ, Goldstein RF, Goldberg RN, Cotten CM; National Institute of Child Health and Human Development Neonatal Research Network. Use of medications for gastroesophageal reflux at discharge among extremely low birth weight infants. Pediatrics. 2008 Jan;121(1):22-7. doi: 10.1542/peds.2007-0381. PMID 18166553
- [Result] Malloy MH, Onstad L, Wright E. The effect of cesarean delivery on birth outcome in very low birth weight infants. National Institute of Child Health and Human Development Neonatal Research Network. Obstet Gynecol. 1991 Apr;77(4):498-503. PMID 2002969
- [Result] Morris BH, Gard CC, Kennedy K; NICHD Neonatal Research Network. Rehospitalization of extremely low birth weight (ELBW) infants: are there racial/ethnic disparities? J Perinatol. 2005 Oct;25(10):656-63. doi: 10.1038/sj.jp.7211361. PMID 16107873
- [Result] Oh W, Tyson JE, Fanaroff AA, Vohr BR, Perritt R, Stoll BJ, Ehrenkranz RA, Carlo WA, Shankaran S, Poole K, Wright LL; National Institute of Child Health and Human Development Neonatal Research Network. Association between peak serum bilirubin and neurodevelopmental outcomes in extremely low birth weight infants. Pediatrics. 2003 Oct;112(4):773-9. doi: 10.1542/peds.112.4.773. PMID 14523165
- [Result] Shankaran S, Bauer CR, Bain R, Wright LL, Zachary J. Prenatal and perinatal risk and protective factors for neonatal intracranial hemorrhage. National Institute of Child Health and Human Development Neonatal Research Network. Arch Pediatr Adolesc Med. 1996 May;150(5):491-7. doi: 10.1001/archpedi.1996.02170300045009. PMID 8620230
- [Result] Shankaran S, Bauer CR, Bain R, Wright LL, Zachary J. Relationship between antenatal steroid administration and grades III and IV intracranial hemorrhage in low birth weight infants. The NICHD Neonatal Research Network. Am J Obstet Gynecol. 1995 Jul;173(1):305-12. doi: 10.1016/0002-9378(95)90219-8. No abstract available. PMID 7631710
- [Result] Shankaran S, Johnson Y, Langer JC, Vohr BR, Fanaroff AA, Wright LL, Poole WK. Outcome of extremely-low-birth-weight infants at highest risk: gestational age < or =24 weeks, birth weight < or =750 g, and 1-minute Apgar < or =3. Am J Obstet Gynecol. 2004 Oct;191(4):1084-91. doi: 10.1016/j.ajog.2004.05.032. PMID 15507925
- [Result] Shankaran S, Fanaroff AA, Wright LL, Stevenson DK, Donovan EF, Ehrenkranz RA, Langer JC, Korones SB, Stoll BJ, Tyson JE, Bauer CR, Lemons JA, Oh W, Papile LA. Risk factors for early death among extremely low-birth-weight infants. Am J Obstet Gynecol. 2002 Apr;186(4):796-802. doi: 10.1067/mob.2002.121652. PMID 11967510
- [Result] St John EB, Carlo WA. Respiratory distress syndrome in VLBW infants: changes in management and outcomes observed by the NICHD Neonatal Research Network. Semin Perinatol. 2003 Aug;27(4):288-92. doi: 10.1016/s0146-0005(03)00056-9. PMID 14510319
- [Result] Stephens BE, Bann CM, Poole WK, Vohr BR. NEURODEVELOPMENTAL IMPAIRMENT: PREDICTORS OF ITS IMPACT ON THE FAMILIES OF EXTREMELY LOW BIRTH WEIGHT INFANTS AT 18 MONTHS. Infant Ment Health J. 2008 Nov 1;29(6):570-587. doi: 10.1002/imhj.20196. PMID 19779585
- [Result] Stevenson DK, Verter J, Fanaroff AA, Oh W, Ehrenkranz RA, Shankaran S, Donovan EF, Wright LL, Lemons JA, Tyson JE, Korones SB, Bauer CR, Stoll BJ, Papile LA. Sex differences in outcomes of very low birthweight infants: the newborn male disadvantage. Arch Dis Child Fetal Neonatal Ed. 2000 Nov;83(3):F182-5. doi: 10.1136/fn.83.3.f182. PMID 11040165
- [Result] Stevenson DK, Wright LL, Lemons JA, Oh W, Korones SB, Papile LA, Bauer CR, Stoll BJ, Tyson JE, Shankaran S, Fanaroff AA, Donovan EF, Ehrenkranz RA, Verter J. Very low birth weight outcomes of the National Institute of Child Health and Human Development Neonatal Research Network, January 1993 through December 1994. Am J Obstet Gynecol. 1998 Dec;179(6 Pt 1):1632-9. doi: 10.1016/s0002-9378(98)70037-7. PMID 9855609
- [Result] Stoll BJ, Gordon T, Korones SB, Shankaran S, Tyson JE, Bauer CR, Fanaroff AA, Lemons JA, Donovan EF, Oh W, Stevenson DK, Ehrenkranz RA, Papile LA, Verter J, Wright LL. Early-onset sepsis in very low birth weight neonates: a report from the National Institute of Child Health and Human Development Neonatal Research Network. J Pediatr. 1996 Jul;129(1):72-80. doi: 10.1016/s0022-3476(96)70192-0. PMID 8757565
- [Result] Stoll BJ, Gordon T, Korones SB, Shankaran S, Tyson JE, Bauer CR, Fanaroff AA, Lemons JA, Donovan EF, Oh W, Stevenson DK, Ehrenkranz RA, Papile LA, Verter J, Wright LL. Late-onset sepsis in very low birth weight neonates: a report from the National Institute of Child Health and Human Development Neonatal Research Network. J Pediatr. 1996 Jul;129(1):63-71. doi: 10.1016/s0022-3476(96)70191-9. PMID 8757564
- [Result] Stoll BJ, Hansen N. Infections in VLBW infants: studies from the NICHD Neonatal Research Network. Semin Perinatol. 2003 Aug;27(4):293-301. doi: 10.1016/s0146-0005(03)00046-6. PMID 14510320
- [Result] Stoll BJ, Hansen N, Fanaroff AA, Lemons JA. Enterobacter sakazakii is a rare cause of neonatal septicemia or meningitis in VLBW infants. J Pediatr. 2004 Jun;144(6):821-3. doi: 10.1016/j.jpeds.2004.02.045. PMID 15192634
- [Result] Stoll BJ, Hansen N, Fanaroff AA, Wright LL, Carlo WA, Ehrenkranz RA, Lemons JA, Donovan EF, Stark AR, Tyson JE, Oh W, Bauer CR, Korones SB, Shankaran S, Laptook AR, Stevenson DK, Papile LA, Poole WK. To tap or not to tap: high likelihood of meningitis without sepsis among very low birth weight infants. Pediatrics. 2004 May;113(5):1181-6. doi: 10.1542/peds.113.5.1181. PMID 15121927
- [Result] Stoll BJ, Hansen N, Fanaroff AA, Wright LL, Carlo WA, Ehrenkranz RA, Lemons JA, Donovan EF, Stark AR, Tyson JE, Oh W, Bauer CR, Korones SB, Shankaran S, Laptook AR, Stevenson DK, Papile LA, Poole WK. Changes in pathogens causing early-onset sepsis in very-low-birth-weight infants. N Engl J Med. 2002 Jul 25;347(4):240-7. doi: 10.1056/NEJMoa012657. PMID 12140299
- [Result] Stoll BJ, Hansen N, Fanaroff AA, Wright LL, Carlo WA, Ehrenkranz RA, Lemons JA, Donovan EF, Stark AR, Tyson JE, Oh W, Bauer CR, Korones SB, Shankaran S, Laptook AR, Stevenson DK, Papile LA, Poole WK. Late-onset sepsis in very low birth weight neonates: the experience of the NICHD Neonatal Research Network. Pediatrics. 2002 Aug;110(2 Pt 1):285-91. doi: 10.1542/peds.110.2.285. PMID 12165580
- [Result] Stoll BJ, Hansen NI, Higgins RD, Fanaroff AA, Duara S, Goldberg R, Laptook A, Walsh M, Oh W, Hale E; National Institute of Child Health and Human Development. Very low birth weight preterm infants with early onset neonatal sepsis: the predominance of gram-negative infections continues in the National Institute of Child Health and Human Development Neonatal Research Network, 2002-2003. Pediatr Infect Dis J. 2005 Jul;24(7):635-9. doi: 10.1097/01.inf.0000168749.82105.64. PMID 15999007
- [Result] Stoll BJ, Hansen NI, Adams-Chapman I, Fanaroff AA, Hintz SR, Vohr B, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental and growth impairment among extremely low-birth-weight infants with neonatal infection. JAMA. 2004 Nov 17;292(19):2357-65. doi: 10.1001/jama.292.19.2357. PMID 15547163
- [Result] Tyson JE, Younes N, Verter J, Wright LL. Viability, morbidity, and resource use among newborns of 501- to 800-g birth weight. National Institute of Child Health and Human Development Neonatal Research Network. JAMA. 1996 Nov 27;276(20):1645-51. PMID 8922450
- [Result] Tyson JE, Parikh NA, Langer J, Green C, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Intensive care for extreme prematurity--moving beyond gestational age. N Engl J Med. 2008 Apr 17;358(16):1672-81. doi: 10.1056/NEJMoa073059. PMID 18420500
- [Result] Uauy RD, Fanaroff AA, Korones SB, Phillips EA, Phillips JB, Wright LL. Necrotizing enterocolitis in very low birth weight infants: biodemographic and clinical correlates. National Institute of Child Health and Human Development Neonatal Research Network. J Pediatr. 1991 Oct;119(4):630-8. doi: 10.1016/s0022-3476(05)82418-7. PMID 1919897
- [Result] Vohr BR, Msall ME, Wilson D, Wright LL, McDonald S, Poole WK. Spectrum of gross motor function in extremely low birth weight children with cerebral palsy at 18 months of age. Pediatrics. 2005 Jul;116(1):123-9. doi: 10.1542/peds.2004-1810. PMID 15995042
- [Result] Vohr BR, O'Shea M, Wright LL. Longitudinal multicenter follow-up of high-risk infants: why, who, when, and what to assess. Semin Perinatol. 2003 Aug;27(4):333-42. doi: 10.1016/s0146-0005(03)00045-4. PMID 14510324
- [Result] Vohr BR, Wright LL, Dusick AM, Mele L, Verter J, Steichen JJ, Simon NP, Wilson DC, Broyles S, Bauer CR, Delaney-Black V, Yolton KA, Fleisher BE, Papile LA, Kaplan MD. Neurodevelopmental and functional outcomes of extremely low birth weight infants in the National Institute of Child Health and Human Development Neonatal Research Network, 1993-1994. Pediatrics. 2000 Jun;105(6):1216-26. doi: 10.1542/peds.105.6.1216. PMID 10835060
- [Result] Vohr BR, Wright LL, Poole WK, McDonald SA. Neurodevelopmental outcomes of extremely low birth weight infants <32 weeks' gestation between 1993 and 1998. Pediatrics. 2005 Sep;116(3):635-43. doi: 10.1542/peds.2004-2247. PMID 16143580
- [Result] Vohr BR, Tyson JE, Wright LL, Perritt RL, Li L, Poole WK; NICHD Neonatal Research Network. Maternal age, multiple birth, and extremely low birth weight infants. J Pediatr. 2009 Apr;154(4):498-503.e2. doi: 10.1016/j.jpeds.2008.10.044. Epub 2008 Dec 25. PMID 19111322
- [Result] Vohr BR, Wright LL, Dusick AM, Perritt R, Poole WK, Tyson JE, Steichen JJ, Bauer CR, Wilson-Costello DE, Mayes LC; Neonatal Research Network. Center differences and outcomes of extremely low birth weight infants. Pediatrics. 2004 Apr;113(4):781-9. doi: 10.1542/peds.113.4.781. PMID 15060228
- [Result] Wadhawan R, Oh W, Perritt R, Laptook AR, Poole K, Wright LL, Fanaroff AA, Duara S, Stoll BJ, Goldberg R. Association between early postnatal weight loss and death or BPD in small and appropriate for gestational age extremely low-birth-weight infants. J Perinatol. 2007 Jun;27(6):359-64. doi: 10.1038/sj.jp.7211751. Epub 2007 Apr 19. PMID 17443198
- [Result] Wadhawan R, Oh W, Perritt RL, McDonald SA, Das A, Poole WK, Vohr BR, Higgins RD. Twin gestation and neurodevelopmental outcome in extremely low birth weight infants. Pediatrics. 2009 Feb;123(2):e220-7. doi: 10.1542/peds.2008-1126. Epub 2009 Jan 12. PMID 19139085
- [Result] Wadhawan R, Vohr BR, Fanaroff AA, Perritt RL, Duara S, Stoll BJ, Goldberg R, Laptook A, Poole K, Wright LL, Oh W. Does labor influence neonatal and neurodevelopmental outcomes of extremely-low-birth-weight infants who are born by cesarean delivery? Am J Obstet Gynecol. 2003 Aug;189(2):501-6. doi: 10.1067/s0002-9378(03)00360-0. PMID 14520225
- [Result] Walden RV, Taylor SC, Hansen NI, Poole WK, Stoll BJ, Abuelo D, Vohr BR; National Institute of Child Health and Human Development Neonatal Research Network. Major congenital anomalies place extremely low birth weight infants at higher risk for poor growth and developmental outcomes. Pediatrics. 2007 Dec;120(6):e1512-9. doi: 10.1542/peds.2007-0354. Epub 2007 Nov 5. PMID 17984212
- [Result] Walsh MC, Morris BH, Wrage LA, Vohr BR, Poole WK, Tyson JE, Wright LL, Ehrenkranz RA, Stoll BJ, Fanaroff AA; National Institutes of Child Health and Human Development Neonatal Research Network. Extremely low birthweight neonates with protracted ventilation: mortality and 18-month neurodevelopmental outcomes. J Pediatr. 2005 Jun;146(6):798-804. doi: 10.1016/j.jpeds.2005.01.047. PMID 15973322
- [Result] Walsh MC, Yao Q, Horbar JD, Carpenter JH, Lee SK, Ohlsson A. Changes in the use of postnatal steroids for bronchopulmonary dysplasia in 3 large neonatal networks. Pediatrics. 2006 Nov;118(5):e1328-35. doi: 10.1542/peds.2006-0359. PMID 17079534
- [Result] Wright LL, Horbar JD, Gunkel H, Verter J, Younes N, Andrews EB, Long W. Evidence from multicenter networks on the current use and effectiveness of antenatal corticosteroids in low birth weight infants. Am J Obstet Gynecol. 1995 Jul;173(1):263-9. doi: 10.1016/0002-9378(95)90211-2. No abstract available. PMID 7631701
- [Result] Wright LL, Verter J, Younes N, Stevenson D, Fanaroff AA, Shankaran S, Ehrenkranz RA, Donovan EF. Antenatal corticosteroid administration and neonatal outcome in very low birth weight infants: the NICHD Neonatal Research Network. Am J Obstet Gynecol. 1995 Jul;173(1):269-74. doi: 10.1016/0002-9378(95)90212-0. No abstract available. PMID 7631702
- [Result] Wright LL; Papile LA. U.S. neonatal databases: methods and uses. Semin Neonatal 1997;2:159-69. (ancillary publication).
- [Result] Ambalavanan N, Carlo WA, Tyson JE, Langer JC, Walsh MC, Parikh NA, Das A, Van Meurs KP, Shankaran S, Stoll BJ, Higgins RD; Generic Database; Subcommittees of the Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Outcome trajectories in extremely preterm infants. Pediatrics. 2012 Jul;130(1):e115-25. doi: 10.1542/peds.2011-3693. Epub 2012 Jun 11. PMID 22689874
- [Derived] Dorner RA, Li L, Lemmon ME, Zangeneh SZ, Das A, Discenza DA, Mancini T, Vaucher Y, Wyckoff MH, Hintz S, DeMauro SB, Carlo WA, Gustafson KE, Katheria A; Eunice Kennedy Schriver National Institute of Child Health and Human Development Neonatal Research Network. Inpatient morbidities and medical technology use at 2 years among extremely preterm infants. Pediatr Res. 2025 Dec 16. doi: 10.1038/s41390-025-04671-0. Online ahead of print. PMID 41402645
- [Derived] Messick EA, Saha S, Slaughter JL, Kielt MJ, Benninger KL, Bell EF, Stoll BJ, Puopolo KM, Mukhopadhyay S, Flannery DD, Wyckoff MH, Cotten CM, Patel RM, Laptook AR, Grisby C, Das A, Walsh MC, Sanchez PJ; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Maternal Coronavirus Disease 2019 Test Positivity and Neonatal Intensive Care Unit Outcomes for Infants Born Extremely Preterm. J Pediatr. 2026 Jan;288:114840. doi: 10.1016/j.jpeds.2025.114840. Epub 2025 Sep 26. PMID 41016465
- [Derived] Kaluarachchi DC, Chock VY, Do BT, Rysavy MA, Sankar MN, Laughon MM, Backes CH, Colaizy TT, Bell EF, McNamara PJ, Hintz SR, Natarajan G. Comparison of neurodevelopmental outcomes of extremely preterm infants undergoing trans-catheter closure of the patent ductus arteriosus compared to surgical ligation. J Perinatol. 2025 Sep 23:10.1038/s41372-025-02417-8. doi: 10.1038/s41372-025-02417-8. Online ahead of print. PMID 40987835
- [Derived] Brumbaugh JE, Bann CM, Bell EF, Travers CP, Vohr BR, McGowan EC, Harmon HM, Carlo WA, Hintz SR, Duncan AF; Eunice Kennedy Shriver NICHD Neonatal Research Network. The Relationship Between Hispanic Ethnicity and Outcomes for Infants Born Extremely Preterm. J Pediatr. 2025 Apr;279:114474. doi: 10.1016/j.jpeds.2025.114474. Epub 2025 Jan 23. PMID 39855622
- [Derived] Kaluarachchi DC, Rysavy MA, Do BT, Chock VY, Laughon MM, Backes CH, Colaizy TT, Bell EF, McNamara PJ. Changes in Patent Ductus Arteriosus Management and Outcomes in Infants Born at 26-28 Weeks' Gestation. J Pediatr. 2025 Apr;279:114456. doi: 10.1016/j.jpeds.2024.114456. Epub 2024 Dec 26. PMID 39732160
- [Derived] Dorner RA, Li L, DeMauro SB, Schmidt B, Zangeneh SZ, Vaucher Y, Wyckoff MH, Hintz S, Carlo WA, Gustafson KE, Das A, Katheria A; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Association of a Count of Inpatient Morbidities with 2-Year Outcomes among Infants Born Extremely Preterm. J Pediatr. 2025 Mar;278:114428. doi: 10.1016/j.jpeds.2024.114428. Epub 2024 Dec 4. PMID 39643110
- [Derived] Honan BM, McDonald SA, Travers CP, Shukla VV, Ambalavanan N, Cotten CM, Jain VG, Arnold HE, Parikh NA, Tyson JE, Hintz SR, Walker SA, Gantz MG, Das A, Carlo WA. Cerebral injury and retinopathy as risk factors for blindness in extremely preterm infants. Arch Dis Child Fetal Neonatal Ed. 2025 Apr 17;110(3):253-260. doi: 10.1136/archdischild-2024-327707. PMID 39332892
- [Derived] Salas AA, Carlo WA, Bann CM, Bell EF, Colaizy TT, Younge N, Peralta M, Ambalavanan N, Poindexter BB; Eunice Kennedy Shriver NICHD Neonatal Research Network. Risk Assessment of Cognitive Impairment at 2 Years of Age in Infants Born Extremely Preterm Using the INTERGROWTH-21st Growth Standards. J Pediatr. 2024 Dec;275:114239. doi: 10.1016/j.jpeds.2024.114239. Epub 2024 Aug 19. PMID 39168179
- [Derived] Aleem S, Do BT, Gantz MG, Hibbs AM, Jensen EA, Cotten CM, Malcolm WF, Jobe AH, Greenberg RG; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. The association of the room air challenge with long-term outcomes in extremely preterm infants. J Perinatol. 2024 Sep;44(9):1300-1306. doi: 10.1038/s41372-024-02074-3. Epub 2024 Aug 3. PMID 39095524
- [Derived] Shukla VV, Carper BA, Ambalavanan N, Rysavy MA, Bell EF, Das A, Patel RM, D'Angio CT, Watterberg KL, Cotten CM, Merhar SL, Wyckoff MH, Sanchez PJ, Kumbhat N, Carlo WA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Social distancing and extremely preterm births in the initial COVID-19 pandemic period. J Perinatol. 2024 Jul;44(7):1050-1057. doi: 10.1038/s41372-024-01898-3. Epub 2024 Feb 22. PMID 38388715
- [Derived] Green CE, Tyson JE, Heyne RJ, Hintz SR, Vohr BR, Bann CM, Das A, Bell EF, Debsareea SB, Stephens E, Gantz MG, Petrie Huitema CM, Johnson KJ, Watterberg KL, Mosquera R, Peralta-Carcelen M, Wilson-Costello DE, Colaizy TT, Maitre NL, Merhar SL, Adams-Chapman I, Fuller J, Hartley-McAndrew ME, Malcolm WF, Winter S, Duncan AF, Myer GJ, Kicklighter SD, Wyckoff MH, DeMauro SB, Hibbs AM, Stoll BJ, Carlo WA, Van Meurs KP, Rysavy MA, Patel RM, Sanchez PJ, Laptook AR, Cotten CM, D'Angio CT, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Use of term reference infants in assessing the developmental outcome of extremely preterm infants: lessons learned in a multicenter study. J Perinatol. 2023 Nov;43(11):1398-1405. doi: 10.1038/s41372-023-01729-x. Epub 2023 Aug 4. PMID 37542155
- [Derived] Kole-White MB, Saha S, Werner EF, Chawla S, Keszler M, McGowan EC, Wyckoff MH, Laptook AR; Generic Database Subcommittee of the Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Maternal hypertensive disorders and survival without major morbidities among extremely low gestation newborns. J Perinatol. 2023 Apr;43(4):430-436. doi: 10.1038/s41372-023-01631-6. Epub 2023 Feb 22. PMID 36813902
- [Derived] Jensen EA, Laughon MM, DeMauro SB, Cotten CM, Do B, Carlo WA, Watterberg KL. Contributions of the NICHD neonatal research network to the diagnosis, prevention, and treatment of bronchopulmonary dysplasia. Semin Perinatol. 2022 Nov;46(7):151638. doi: 10.1016/j.semperi.2022.151638. Epub 2022 Jun 10. PMID 36085059
- [Derived] Kilbride HW, Vohr BR, McGowan EM, Peralta-Carcelen M, Stringer K, Das A, Archer SW, Hintz SR. Early neurodevelopmental follow-up in the NICHD neonatal research network: Advancing neonatal care and outcomes, opportunities for the future. Semin Perinatol. 2022 Nov;46(7):151642. doi: 10.1016/j.semperi.2022.151642. Epub 2022 Jun 10. PMID 35842320
- [Derived] Bell EF, Stoll BJ, Hansen NI, Wyckoff MH, Walsh MC, Sanchez PJ, Rysavy MA, Gabrio JH, Archer SW, Das A, Higgins RD. Contributions of the NICHD neonatal research network's generic database to documenting and advancing the outcomes of extremely preterm infants. Semin Perinatol. 2022 Nov;46(7):151635. doi: 10.1016/j.semperi.2022.151635. Epub 2022 Jun 10. PMID 35835615
- [Derived] Greenberg RG, McDonald SA, Laughon MM, Tanaka D, Jensen E, Van Meurs K, Eichenwald E, Brumbaugh JE, Duncan AF, Walsh M, Das A, Cotten CM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Online clinical tool to estimate risk of bronchopulmonary dysplasia in extremely preterm infants. Arch Dis Child Fetal Neonatal Ed. 2022 Jun 21:fetalneonatal-2021-323573. doi: 10.1136/archdischild-2021-323573. Online ahead of print. PMID 35728925
- [Derived] Puopolo KM, Mukhopadhyay S, Hansen NI, Flannery DD, Greenberg RG, Sanchez PJ, Bell EF, DeMauro SB, Wyckoff MH, Eichenwald EC, Stoll BJ. Group B Streptococcus Infection in Extremely Preterm Neonates and Neurodevelopmental Outcomes at 2 Years. Clin Infect Dis. 2022 Oct 12;75(8):1405-1415. doi: 10.1093/cid/ciac222. PMID 35323895
- [Derived] Gentle SJ, Carper B, Laughon MM, Jensen EA, Williams A, Travers CP, Ambalavanan N, Lal CV, Carlo WA. Duration of noninvasive respiratory support and risk for bronchopulmonary dysplasia or death. J Perinatol. 2022 Apr;42(4):454-460. doi: 10.1038/s41372-021-01269-2. Epub 2022 Jan 15. PMID 35034096
- [Derived] Kumbhat N, Eggleston B, Davis AS, DeMauro SB, Van Meurs KP, Foglia EE, Lakshminrusimha S, Walsh MC, Watterberg KL, Wyckoff MH, Das A, Handley SC; Generic Database Subcommittee of the National Institute of Child Health and Human Development Neonatal Research Network. Umbilical Cord Milking vs Delayed Cord Clamping and Associations with In-Hospital Outcomes among Extremely Premature Infants. J Pediatr. 2021 May;232:87-94.e4. doi: 10.1016/j.jpeds.2020.12.072. Epub 2021 Jan 5. PMID 33417919
- [Derived] Chandrasekharan P, Lakshminrusimha S, Chowdhury D, Van Meurs K, Keszler M, Kirpalani H, Das A, Walsh MC, McGowan EC, Higgins RD; NRN STEERING COMMITTEE. Early Hypoxic Respiratory Failure in Extreme Prematurity: Mortality and Neurodevelopmental Outcomes. Pediatrics. 2020 Oct;146(4):e20193318. doi: 10.1542/peds.2019-3318. Epub 2020 Sep 17. PMID 32943536
- [Derived] Shankaran S, Bajaj M, Natarajan G, Saha S, Pappas A, Davis AS, Hintz SR, Adams-Chapman I, Das A, Bell EF, Stoll BJ, Walsh MC, Laptook AR, Carlo WA, Van Meurs KP, Sanchez PJ, Ball MB, Hale EC, Seabrook R, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Outcomes Following Post-Hemorrhagic Ventricular Dilatation among Infants of Extremely Low Gestational Age. J Pediatr. 2020 Nov;226:36-44.e3. doi: 10.1016/j.jpeds.2020.07.080. Epub 2020 Jul 30. PMID 32739261
- [Derived] Kumbhat N, Eggleston B, Davis AS, Van Meurs KP, DeMauro SB, Foglia EE, Lakshminrusimha S, Walsh MC, Watterberg KL, Wyckoff MH, Das A, Handley SC; Generic Database Subcommittee of the NICHD Neonatal Research Network; undefined. Placental transfusion and short-term outcomes among extremely preterm infants. Arch Dis Child Fetal Neonatal Ed. 2021 Jan;106(1):62-68. doi: 10.1136/archdischild-2019-318710. Epub 2020 Jul 30. PMID 32732380
- [Derived] Gentle SJ, Carlo WA, Tan S, Gargano M, Ambalavanan N, Chawla S, Bell EF, Bann CM, Hintz SR, Heyne RJ, Tita A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Neonatal Research Network. Association of Antenatal Corticosteroids and Magnesium Sulfate Therapy With Neurodevelopmental Outcome in Extremely Preterm Children. Obstet Gynecol. 2020 Jun;135(6):1377-1386. doi: 10.1097/AOG.0000000000003882. PMID 32459430
- [Derived] Warren MG, Do B, Das A, Smith PB, Adams-Chapman I, Jadcherla S, Jensen EA, Goldstein RF, Goldberg RN, Cotten CM, Bell EF, Malcolm WF; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Gastrostomy Tube Feeding in Extremely Low Birthweight Infants: Frequency, Associated Comorbidities, and Long-term Outcomes. J Pediatr. 2019 Nov;214:41-46.e5. doi: 10.1016/j.jpeds.2019.06.066. Epub 2019 Aug 16. PMID 31427096
- [Derived] DeMauro SB, Jensen EA, Bann CM, Bell EF, Hibbs AM, Hintz SR, Lorch SA. Home Oxygen and 2-Year Outcomes of Preterm Infants With Bronchopulmonary Dysplasia. Pediatrics. 2019 May;143(5):e20182956. doi: 10.1542/peds.2018-2956. Epub 2019 Apr 11. PMID 30975699
- [Derived] Rysavy MA, Bell EF, Iams JD, Carlo WA, Li L, Mercer BM, Hintz SR, Stoll BJ, Vohr BR, Shankaran S, Walsh MC, Brumbaugh JE, Colaizy TT, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Discordance in Antenatal Corticosteroid Use and Resuscitation Following Extremely Preterm Birth. J Pediatr. 2019 May;208:156-162.e5. doi: 10.1016/j.jpeds.2018.12.063. Epub 2019 Feb 6. PMID 30738658
- [Derived] Duncan AF, Bann CM, Dempsey AG, Adams-Chapman I, Heyne R, Hintz SR; Eunice Kennedy Shriver National Institute of Child Health and Development Neonatal Research Network. Neuroimaging and Bayley-III correlates of early hand function in extremely preterm children. J Perinatol. 2019 Mar;39(3):488-496. doi: 10.1038/s41372-019-0314-0. Epub 2019 Jan 28. PMID 30692613
- [Derived] Lowe JR, Fuller JF, Do BT, Vohr BR, Das A, Hintz SR, Watterberg KL, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health; Human Development Neonatal Research Network. Behavioral problems are associated with cognitive and language scores in toddlers born extremely preterm. Early Hum Dev. 2019 Jan;128:48-54. doi: 10.1016/j.earlhumdev.2018.11.007. Epub 2018 Dec 4. PMID 30522091
- [Derived] Duncan AF, Bann CM, Dempsey A, Peralta-Carcelen M, Hintz S; Eunice Kennedy Shriver National Institute of Child Health and Development Neonatal Research Network. Behavioral Deficits at 18-22 Months of Age Are Associated with Early Cerebellar Injury and Cognitive and Language Performance in Children Born Extremely Preterm. J Pediatr. 2019 Jan;204:148-156.e4. doi: 10.1016/j.jpeds.2018.08.059. Epub 2018 Oct 3. PMID 30292492
- [Derived] Vohr BR, Heyne R, Bann CM, Das A, Higgins RD, Hintz SR; Eunice Kennedy Shriver National Institute of Child Health, and Development Neonatal Research Network. Extreme Preterm Infant Rates of Overweight and Obesity at School Age in the SUPPORT Neuroimaging and Neurodevelopmental Outcomes Cohort. J Pediatr. 2018 Sep;200:132-139.e3. doi: 10.1016/j.jpeds.2018.04.073. Epub 2018 May 21. PMID 29793869
- [Derived] Adams-Chapman I, Heyne RJ, DeMauro SB, Duncan AF, Hintz SR, Pappas A, Vohr BR, McDonald SA, Das A, Newman JE, Higgins RD; Follow-Up Study of the Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental Impairment Among Extremely Preterm Infants in the Neonatal Research Network. Pediatrics. 2018 May;141(5):e20173091. doi: 10.1542/peds.2017-3091. Epub 2018 Apr 17. PMID 29666163
- [Derived] Boghossian NS, Do BT, Bell EF, Dagle JM, Brumbaugh JE, Stoll BJ, Vohr BR, Das A, Shankaran S, Sanchez PJ, Wyckoff MH, Bethany Ball M; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Efficacy of pharmacologic closure of patent ductus arteriosus in small-for-gestational-age extremely preterm infants. Early Hum Dev. 2017 Oct;113:10-17. doi: 10.1016/j.earlhumdev.2017.07.011. Epub 2017 Jul 8. PMID 28697406
- [Derived] James J, Munson D, DeMauro SB, Langer JC, Dworetz AR, Natarajan G, Bidegain M, Fortney CA, Seabrook R, Vohr BR, Tyson JE, Bell EF, Poindexter BB, Shankaran S, Higgins RD, Das A, Stoll BJ, Kirpalani H; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Outcomes of Preterm Infants following Discussions about Withdrawal or Withholding of Life Support. J Pediatr. 2017 Nov;190:118-123.e4. doi: 10.1016/j.jpeds.2017.05.056. Epub 2017 Jun 21. PMID 28647272
- [Derived] Jensen EA, Dysart KC, Gantz MG, Carper B, Higgins RD, Keszler M, Laughon MM, Poindexter BB, Stoll BJ, Walsh MC, Schmidt B; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Association between Use of Prophylactic Indomethacin and the Risk for Bronchopulmonary Dysplasia in Extremely Preterm Infants. J Pediatr. 2017 Jul;186:34-40.e2. doi: 10.1016/j.jpeds.2017.02.003. Epub 2017 Feb 28. PMID 28258737
- [Derived] Younge N, Goldstein RF, Bann CM, Hintz SR, Patel RM, Smith PB, Bell EF, Rysavy MA, Duncan AF, Vohr BR, Das A, Goldberg RN, Higgins RD, Cotten CM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Survival and Neurodevelopmental Outcomes among Periviable Infants. N Engl J Med. 2017 Feb 16;376(7):617-628. doi: 10.1056/NEJMoa1605566. PMID 28199816
- [Derived] Boghossian NS, Hansen NI, Bell EF, Brumbaugh JE, Stoll BJ, Laptook AR, Shankaran S, Wyckoff MH, Colaizy TT, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Outcomes of Extremely Preterm Infants Born to Insulin-Dependent Diabetic Mothers. Pediatrics. 2016 Jun;137(6):e20153424. doi: 10.1542/peds.2015-3424. Epub 2016 May 13. PMID 27244849
- [Derived] Stoll BJ, Hansen NI, Bell EF, Walsh MC, Carlo WA, Shankaran S, Laptook AR, Sanchez PJ, Van Meurs KP, Wyckoff M, Das A, Hale EC, Ball MB, Newman NS, Schibler K, Poindexter BB, Kennedy KA, Cotten CM, Watterberg KL, D'Angio CT, DeMauro SB, Truog WE, Devaskar U, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Trends in Care Practices, Morbidity, and Mortality of Extremely Preterm Neonates, 1993-2012. JAMA. 2015 Sep 8;314(10):1039-51. doi: 10.1001/jama.2015.10244. PMID 26348753
- [Derived] LeVan JM, Brion LP, Wrage LA, Gantz MG, Wyckoff MH, Sanchez PJ, Heyne R, Jaleel M, Finer NN, Carlo WA, Das A, Stoll BJ, Higgins RD; Eunice Kennedy Shriver NICHD Neonatal Research Network. Change in practice after the Surfactant, Positive Pressure and Oxygenation Randomised Trial. Arch Dis Child Fetal Neonatal Ed. 2014 Sep;99(5):F386-90. doi: 10.1136/archdischild-2014-306057. Epub 2014 May 29. PMID 24876196
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/
- See also: NICHD Pregnancy & Perinatology Branch — https://www.nichd.nih.gov/about/org/der/branches/ppb